CLINICAL TRIAL: NCT06062537
Title: Analysis of Effectiveness and Safety of Teclistamab in Relapsed and Refractory Multiple Myeloma Patients: a Collaborative Janssen - IFM Study IFM 2023-01: TEC-CARE
Brief Title: Analysis of Effectiveness and Safety of Teclistamab in Relapsed and Refractory Multiple Myeloma Patients
Acronym: TEC-CARE
Status: Active, not recruiting | Type: Observational
Sponsor: Intergroupe Francophone du Myelome (Network)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: IFM 2023-01
Record Dates: First submitted 2023-09-22; First posted 2023-10-02 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Multiple Myeloma
Keywords: teclistamab; refractory multiple myeloma; real word evidence study
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
200 adult patients with multiple myeloma receiving teclistamb will be included. Effectiveness, safety, and condition of use of teclistamab in early access program (post-MA) will be assessed. Primary objective is the evaluation of overall response rate (ORR) of teclistamab according to IMWG criteria.

This is a multicenter, prospective, observational study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years) with multiple myeloma who will receive at least one dose of teclistamab (first dose of the step-up dose)

Exclusion Criteria:

* Patients alive at the start of the study who did not receive study information or who objected to the collection of data
* Patients who received teclistamab as part of an interventional clinical trial
* Patients who are initiating teclistamab as part of a current interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: French adult patient relapsed and refractory multiple myeloma receving teclistamab
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
overall response rate (ORR) of teclistamab according to IMWG criteria | 6 months
  ORR is defined as the proportion of subjects who achieve a PR or better according to IMWG criteria.
overall response rate (ORR) of teclistamab according to IMWG criteria | 24 months
  ORR is defined as the proportion of subjects who achieve a PR or better according to IMWG criteria.

SECONDARY OUTCOMES:
Effectiveness of teclistamab | 24 months
  Progression Free Survival 1 and 2 (PFS)
Effectiveness of teclistamab | 24 months
  Overall survival (OS)
Effectiveness of teclistamab | 24 months
  Duration of overall response (DOR)
Effectiveness of teclistamab | 24 months
  Response rate (sCR, CR, VGPR, PR)
Effectiveness of teclistamab | 24 months
  Time to best response
Effectiveness of teclistamab | 24 months
  Time to next treatment (TTNT)
Effectiveness of teclistamab | 24 months
  Time to discontinuation (TTD)
Adverse events of interest | 24 months
  ICANS, CSR and infections
Conditions of use | 1 month
  Patients' profiles (demographics characteristics and medical history)
  - Injection facilities and schedules during step-up dosing phase
Conditions of use | 24 months
  Patients' profiles (demographics characteristics and medical history)
  - Injection facilities and schedules during follow up phase

CONTACTS AND LOCATIONS:
Locations (31):
- France (31):
  - CHU Amiens Picardie, Amiens
  - CH d'ANNECY, Annecy
  - Centre hospitalier d'Argenteuil, Argenteuil
  - Hopital de la cote Basque, Bayonne
  - CHU de Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - Centre hospitalier de Brive-la-Gaillarde, Brive-la-Gaillarde
  - CHU CAEN, Caen
  - Centre hospitalier Métropole de Savoie, Chambéry
  - CHU Clermont-Ferrand Site Estaing, Clermont-Ferrand
  - CHU Henri Mondor, Créteil
  - Chu Dijon, Dijon
  - CH Dunkerque, Dunkirk
  - CHU de Lille, Lille
  - Groupe hospitalier Bretagne Sud, Lorient
  - Institut Paoli Calmette, Marseille
  - CH de METZ, Metz
  - CHU Saint-Eloi - CHU de Montpellier, Montpellier
  - Chu de Nantes, Nantes
  - CHU de Nice, Nice
  - Hopital Necker, Paris
  - Hopital saint louis, Paris
  - CH Perpignan, Perpignan
  - Hopital Novo, Pontoise
  - Chu de Rennes, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut de Cancérologie Lucien Neuwirth, CHU Saint-Etienne, Saint-Priest-en-Jarez
  - Institut de Cancérologie Strasbourg Europe, Strasbourg
  - CHU Toulouse, Toulouse
  - CHU de Tours, Tours
  - CH Bretagne Atlantique, Vannes